CLINICAL TRIAL: NCT03898219
Title: Hematogenous Osteomyelitis in Childhood Can Relapse Dozens of Years in Adulthood
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0262
Record Dates: First submitted 2017-06-19; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Osteomyelitis; Hematogenous Osteomyelitis Relapse
Keywords: Hematogenous osteomyelitis; relapse; adulthood
MeSH Terms: conditions — Osteomyelitis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To our knowledge, few cases of relapse in adulthood are described in the literature except in patients with sickle cell disease and the epidemiological, clinical, laboratory, radiological features and the management of osteomyelitis relapsing in adulthood are not described. The aim of this retrospective multicentric cohort study : in France is to describe the epidemiological, clinical, laboratory, and radiological features and the management of adult patients who experienced a relapse between 2003-2015 of an acute hematogenous osteomyelitis acquired in the childhood (description of characterization of the period between the first episode of osteomyelitis and the second episode, description of signs of relapse and description of treatments used in the relapse). The data are analysed with non-comparative descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) who presented a relapse between 2003-2015 of a hematogenous osteomyelitis acquired in childhood.
* the time limit between the 2 episodes must be at least 2 years
* antecedent of osteomyelitis before 16 years

Exclusion Criteria:

* inability to give the information to the patient
* patients opposed to the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) who presented a relapse between 2003-2015 of a hematogenous osteomyelitis acquired in childhood.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

PRIMARY OUTCOMES:
Rate of patients having an osteomyelitis | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of the population

SECONDARY OUTCOMES:
rate of bacteria responsible for infection | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  bacterial epidemiology
rate of management with surgery | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of type of surgery
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse, Lyon, France